CLINICAL TRIAL: NCT03309007
Title: A Double-Blind, Placebo-Controlled Trial of Anti-Aging, Pro-Autophagy Effects of Metformin in Adults With Prediabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-214
Record Dates: First submitted 2017-07-07; First posted 2017-10-13 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: PreDiabetes; Aging
Keywords: Autophagy
MeSH Terms: conditions — Prediabetic State | interventions — Metformin; Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: This is a double-blind, approximate placebo-controlled trial of 12 weeks of metformin vs. CaCO3 (Placebo) among adult patients with prediabetes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the study research pharmacy will have access to the randomization list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Metformin started at 500 mg po twice daily (BID), and then titrated up to 1000 mg po q morning (AM) and 500 po q evening (PM) over the course of 1 month, as tolerated.
  Interventions: Drug: Metformin
- Placebo Oral Tablet (Placebo Comparator): Near-identical CaCO3 as a Placebo Oral Tablet will be started at 648 mg po BID, and then titrated up to 1296 mg po q AM and 648 mg po q PM over the course of 1 month, as tolerated.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Metformin — Total daily dose titrated up to 1500 mg po q day over the course of 4 weeks and continued for a total exposure of 12 weeks.
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo Oral Tablet — Total daily dose titrated up to 1944 mg po q day over the course of 4 weeks and continued for a total exposure of 12 weeks.
  Other Names: Calcium Carbonate
  Arms: Placebo Oral Tablet

SUMMARY:
The goal of this pilot and feasibility study is to investigate the effects of a short course of metformin therapy on a surrogate marker of cellular senescence and autophagy among adult patients with prediabetes. The overall hypothesis is that metformin will have beneficial effects on longevity and quality of life by inducing autophagy downstream of activating adenosine monophosphate-activated protein kinase (AMPK) and inhibiting mechanistic target of rapamycin (mTOR) through potential effects of reduced inflammation, reduced degeneration of muscle and tendon tissue, antineoplastic effects, reduced obesity and hyperglycemia, preserved cardiovascular functions, and/or the prevention of neurodegeneration (such as age-associated dementia). This pilot study will address the following aim:

Demonstrate that metformin therapy will increase cellular autophagy as an inverse correlate of aging as measured by increases in Microtubule-associated protein 1A/1B-light chain 3 (LC3) scores.

Hypothesis 1: In addition to beneficial effects on glycemia, body weight, and body composition, metformin therapy exerts beneficial effects on surrogate measures of autophagy and aging.

Primary outcome: Increased levels of LC3 in leukocytes.

DETAILED DESCRIPTION:
Anti-aging medicine is a burgeoning field. Accumulating evidence implicates the cellular process of autophagy as a primary mechanism of normal aging and the diseases associated with it. Autophagy is a process of "cellular recycling" and is known to affect a spectrum of health and disease states associated with aging, including inflammatory disorders, metabolic syndrome, type 2 diabetes, cardiovascular disease, cancer, and neurodegeneration. The dynamics of autophagy are controlled by autophagy-related genes and by one of the central regulators of metabolism, AMPK (the target of metformin). Autophagy also affects stem cells and cellular senescence. When the process of autophagy fails, the result is a state of chronic inflammation and degeneration in many organ systems.

Numerous studies have documented the metabolic benefits conferred by the glucose lowering agent metformin. In animal models, metformin has been shown to increase both lifespan and health-span, and a clinical trial (NCT02432287) is currently ongoing to determine whether this effect translates to humans, with additional investigation into how the medication alters the adult human transcriptome. In vitro studies demonstrate metformin's ability to mitigate aging- and disease-related inflammation, oxidative damage, and diminished autophagy. Additionally, there are numerous cohort, case-control and meta-analysis studies confirming metformin's reduction in cancer-related death via hypothesized activity in the relevant mTOR, human epidermal growth factor receptor 2 (HER2), micro-Ribosomal Nucleic Acid (miRNA) and transcription growth factor alpha (TGF-alpha) pathways and processes. As such, the National Institutes of Health (NIH) has issued an Funding Opportunity Announcement (FOA) parent announcement PA-17-073 (https://grants.nih.gov/grants/guide/pa-files/PA-17-073.html) to solicit additional clinical studies that will evaluate metformin's effects on aging and age-related conditions.

The long term goal of this study is to develop a Phase III study in response to this FOA using leucocyte LC3, transcription factor EB (TFEB) scores, total DNA methylation and galectin-3 to gauge the magnitude of metformin's effects on autophagy and cellular senescence as proxies for aging in adults with prediabetes. This study will provide preliminary data for such a proposal, and it will fill a knowledge gap regarding the use of validated biomarkers in this arena. It will also contribute significantly to the anti-aging literature. The primary objective of this proposal is to validate the autophagy-related experimental design by using leucocyte LC3 as a marker of autophagy and cellular senescence in humans.

Aim: Demonstrate that metformin therapy will increase cellular autophagy as an inverse correlate of aging as measured by increases in LC3 scores.

Hypothesis 1: In addition to beneficial effects on glycemia, body weight, and body composition, metformin therapy exerts beneficial effects on surrogate measures of autophagy and aging.

Primary outcome: Increased levels of LC3.

FUTURE DIRECTIONS Confirmation of improvement in markers of autophagy resulting from treatment with metformin will justify the submission of grant proposals for more definitive clinical trials examining the effect of metformin on actual clinical outcomes (as opposed to surrogate measures) in pursuit of a potential Food and Drug Administration (FDA) indication for metformin as an anti-aging therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults with prediabetes (defined as an A1c of 5.7-6.4%)
* BMI between 27 and 40 kg/m2 (inclusive).

Exclusion Criteria:

* Prior treatment with metformin or other diabetes medications,
* Pregnancy,
* Significant renal dysfunction (Serum Creatinine > 1.3 mg/dl for women, > 1.4 mg/dl for men),
* Severe hepatic dysfunction (aspartate amnotransferease [AST] or alanine aminotransferase [ALT] > 3 times the upper limit of normal),
* Ongoing alcohol or substance abuse,
* Inflammatory bowel disease,
* Ongoing glucocorticoid therapy,
* Or inability to render informed consent.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Burge, MD, Principal Investigator — Professor Medicine, UNM HSC Endocrinology
Locations (1):
- University of New Mexico Clincal & Translational Science Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available for data sharing as is consistent with current NIH guidelines.
Supporting Information: Study Protocol, ICF
Time Frame: After the study is completed and published. The data should be available in perpetuity in the University of New Mexico (UNM) Digital Repository.
Access Criteria: No restrictions.
URL: http://digitalrepository.unm.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin | Placebo Oral Tablet
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Metformin: Metformin 500 mg po BID titrated to 1000 q AM and 500 q PM over one month, as tolerated.
- Placebo Oral Tablet: Placebo (CaCO3) 648 mg po BID titrated to 1296 qAM and 648 q PM over one month, as tolerated.
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo Oral Tablet | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 3 | 7 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.1) | 62.3 (7.4) | 60.8 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total 25 enrolled
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 11 | 12 | 23
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Leucocyte LC3 Score
Description: During the process of autophagy, autophagosomes engulf cytoplasmic components and concomitantly, the cytosolic form of LC3 (LC3-I) is conjugated to phosphatidyl ethanolamine, resulting in the autophagosomal membrane-bound form (LC3-II). LC3-II is a widely used marker to monitor autophagosome formation by quantitation of the number of LC3-labeled puncta (autophagosomes, or "dots") per cell detected by fluorescence microscopy. An increase in LC3 puncta formation denotes an increase in autophagic activity.
Time Frame: Data will be collected at 0 and 12 weeks and analyzed within 8 weeks of sample collection.
Measure: Mean (Standard Deviation); unit: Fold Change (Arbitrary Units)
Arm/Group | Metformin | Placebo Oral Tablet
Number analyzed (Participants) | 13 | 12
Fold Change (Arbitrary Units) | 0.1 (3.4) | -1.8 (3.0)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Metformin | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 1/13 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=13) | Placebo Oral Tablet (N=12)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT03309007/Prot_SAP_002.pdf
  • Informed Consent Form (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT03309007/ICF_006.pdf